CLINICAL TRIAL: NCT06409806
Title: Electrocorticography As a Neurophysiological Marker for Intraoperative Monitoring for Brain Retraction: an IDEAL Stage 1 Study
Brief Title: Electrocorticographic Monitoring of Brain Retraction Injury (EMBRI)
Acronym: EMBRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 310742
Record Dates: First submitted 2024-05-01; First posted 2024-05-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Brain Injury; Neurosurgery; Brain Ischemia
Keywords: Brain retraction
MeSH Terms: conditions — Brain Injuries; Brain Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Other: ECOG Array

INTERVENTIONS:
Other: ECOG Array — The patient will undergo their intracranial neurosurgical procedure as planned, using conventional brain retractors and neurosurgical equipment.
  Standard neuromonitoring (EEG, MEP, SSEP) will be placed after the induction of neuroanaesthesia if indicated. Additional to whatever conventional EMBRI neuromonitoring is used, intraoperatively an ECoG array will be positioned under the retractor by the operating surgeon. Further electrode arrays may be placed on the cortical surface remote from the retractor as needed to establish a reference.
  Typically we anticipate one ECoG array under the retractor blade with a reference array on an area of unretracted brain.

SUMMARY:
A single centre IDEAL Stage 1 feasibility study using novel electrophysiological recording techniques in adult participants undergoing neurosurgery. This is a first in human study, building upon previous preclinical mice experiments.

Participants will undergo their planned neurosurgical procedure as normal. In addition to their standard treatment neurophysiological monitoring including an electrocorticography electrode placed on the brain deep to the retractor will be used to monitor for signs of brain retraction injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 or older undergoing intracranial surgery where it is anticipated fixed brain retraction will be used.

Exclusion Criteria:

* Patients without capacity to give consent at time of recruitment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of integrating the ECoG brain retractor into standard traditional neurosurgical operative workflow. | Over a 28 month period from November 2022 to March 2026
  The primary outcome is to report the feasibility of integrating the ECoG brain retractor into standard traditional neurosurgical operative workflow based upon analysing prospective data including qualitative questionnaires administered to surgeons and scrub nurses, anonymised clinical data, and anonymised electrophysiological data.
  The primary outcome is to produce a descriptive report of the electrophysiological data recorded and the challenges encountered in the delivery of the novel electrophysiological recording for patients undergoing planned neurosurgical procedures at the National Hospital for Neurology and Neurosurgery, London.

SECONDARY OUTCOMES:
Analyse the captured electrophysiological data to investigate any correlation between the electrophysiological signature and duration of retraction. | Over a 28 month period from November 2022 to March 2026
  The secondary objective is to analyse the captured electrophysiological data to investigate any correlation between the electrophysiological signature and duration of retraction. Post-operative clinical data, such as MRI brain scans, can be reviewed to investigate any ischemic events.
  We will perform an initial analysis of the electrophysiological data to see if neurophysiological stigmata of brain retraction injury can be identified, with the operation simultaneous recorded with the operative microscope.

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital Neurology and Neurosurgery, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No